CLINICAL TRIAL: NCT02719925
Title: Effect of One Month of Daily Consumption of Mineral Water Rich in Magnesium on Perceived Stress in Healthy Consumers.
Brief Title: Mineral Water Rich in Magnesium and Perceived Stress in Healthy Consumers
Acronym: STRESSOM15
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: My Goodlife SAS (Industry)
Collaborators: Neptune (Industry)
Responsible Party: Principal Investigator, Sebastien Czernichow, Co founder of MGL, My Goodlife SAS
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MGL-002
Record Dates: First submitted 2016-03-21; First posted 2016-03-25 (Estimated); Last update posted 2018-08-27 (Actual); Status verified 2018-08

CONDITIONS: Magnesium Deficiency; Stress, Psychological
Keywords: magnesium deficiency; stress psycological; sleep duration and quality; mineral water rich in magnesium
MeSH Terms: conditions — Magnesium Deficiency; Stress, Psychological

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mineral water rich in magnesium (Experimental): - 1,5 L per day of mineral water containing 160 mg/L of magnesium
  Interventions: Other: Mg(+)
- Water low in magnesium (Active Comparator): - 1,5 L per day of mineral water containing 50 mg/L of magnesium
  Interventions: Other: Mg(-)

INTERVENTIONS:
Other: Mg(+) — * 1,5 L per day during 30 days
  * No livestyle counseling
  Arms: Mineral water rich in magnesium
Other: Mg(-) — 1,5 L water per day during 30 days No lifestyle counseling
  Arms: Water low in magnesium

SUMMARY:
The goal of clinical trial is to evaluate the effect of one month of consumption of mineral water rich in magnesium or not on perceived stress, duration and quality of sleep in healthy consumers having magnesium daily intakes below the recommended dietary allowance (RDA).

DETAILED DESCRIPTION:
This is a single-center, double-blind, controlled, randomized, 2 parallel-groups clinical trial.

256 healthy volunteers will be recruited for clinical trial if they meet the inclusion and no inclusion criteria.

50% of volunteers (Mg+ group) will drink daily 1,5 L of mineral water rich in magnesium during 30 days

50% of volunteers (Mg- group) will drink daily 1,5 L of water low in magnesium during 30 days

Volunteers in both groups will be equipped with a wristband-connected device allowing recording of duration and quality of sleep.

ELIGIBILITY:
Inclusion Criteria:

* a magnesium daily intakes lower than the recommended dietary allowance (RDA)
* a score at perceived stress scale (PPS) greater than or equal to 25
* BMI > 18 et < 25 kg/m2
* Describing himself as tired for reasons of stress or lack of sleep.
* Do not take any medication likely to act on stress and sleep as anxiolytics, hypnotics, antidepressants, etc.
* Knowing read and write French routinely,
* Possessing an internet connection at home,
* Possessing and knowing how to use a computer or tablet,
* Owning a smartphone,
* Affiliated with a social security scheme
* Not Trust
* Having signed the informed consent letter

Exclusion Criteria:

* Pregnant or breast-feeding or planning an early pregnancy during the study
* Severe chronic condition or type of acute disease: vascular cardio - pulmonary - renal - Hematologic - Liver - endocrine (thyroid) - allergic
* Inability to understand information about the protocol and / or to sign the informed consent

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 256 (Actual)
Dates: Start 2016-07; Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Change from baseline score obtained at PSS | At Day 30
  Difference of score obtained at PSS self-administrated questionnaire at Day 30 and Day 0

SECONDARY OUTCOMES:
Change from baseline score obtained at IPAQ | At Day 30
  Difference of score obtained at IPAQ self-administrated questionnaire at Day 30 and Day 0
Change from baseline mean duration of sleep at Week 4 | At week 4
  Difference of the mean duration of sleep during the week before consumption of water and during the fourth week of consumption of water.
Change from baseline mean quality of sleep recorded at Week 4 | At week 4
  Difference of the mean quality of sleep during the week before consumption of water and during the fourth week of consumption of water.

CONTACTS AND LOCATIONS:
Overall Officials: Karl AUZOU, Study Director — MY GOODLIFE
Locations (1):
- My Goodlife, Paris, Île-de-France Region, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] McCabe D, Colbeck M. The effectiveness of essential fatty acid, B vitamin, Vitamin C, magnesium and zinc supplementation for managing stress in women: a systematic review protocol. JBI Database System Rev Implement Rep. 2015 Aug 14;13(7):104-18. doi: 10.11124/jbisrir-2015-2298. No abstract available. PMID 26455850
- [Background] Endoh K, Kuriki K, Kasezawa N, Tohyama K, Goda T. Interactions between psychological stress and drinking status in relation to diet among middle-aged men and women: a large-scale cross-sectional study in Japan. J Nutr Sci Vitaminol (Tokyo). 2015;61(1):64-72. doi: 10.3177/jnsv.61.64. PMID 26027597
- [Background] Vanaelst B, Michels N, Huybrechts I, Clays E, Florez MR, Balcaen L, Resano M, Aramendia M, Vanhaecke F, Rivet N, Raul JS, Lanfer A, De Henauw S. Cross-sectional relationship between chronic stress and mineral concentrations in hair of elementary school girls. Biol Trace Elem Res. 2013 Jun;153(1-3):41-9. doi: 10.1007/s12011-013-9647-2. Epub 2013 Apr 2. PMID 23546894
- [Background] Sartori SB, Whittle N, Hetzenauer A, Singewald N. Magnesium deficiency induces anxiety and HPA axis dysregulation: modulation by therapeutic drug treatment. Neuropharmacology. 2012 Jan;62(1):304-12. doi: 10.1016/j.neuropharm.2011.07.027. Epub 2011 Aug 4. PMID 21835188
- [Background] Grases G, Perez-Castello JA, Sanchis P, Casero A, Perello J, Isern B, Rigo E, Grases F. Anxiety and stress among science students. Study of calcium and magnesium alterations. Magnes Res. 2006 Jun;19(2):102-6. PMID 16955721